CLINICAL TRIAL: NCT00952198
Title: A Safety Study of ARRY-403 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ARRAY-403-102
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ARRY-403

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARRY-403 (Experimental)
  Interventions: Drug: ARRY-403, glucokinase activator; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-403, glucokinase activator; oral — multiple dose, escalating
  Arms: ARRY-403
Drug: Placebo; oral — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 study, involving a 10-day dosing period, designed to test the safety of investigational study drug ARRY-403 (as monotherapy or in addition to stable metformin therapy) in patients with Type 2 diabetes. Approximately 128 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female (females must be of non-childbearing potential), between the ages of 18 and 70 years, inclusive.
* Diagnosis of Type 2 diabetes.
* Fasted C-peptide value ≥ 0.8 ng/mL.
* HbA1c ≥ 6.5% and ≤ 10.0% for monotherapy cohorts (study drug only) or HbA1c ≥ 7.5% and ≤ 10.0% for combination cohorts (study drug and on a stable regimen of metformin monotherapy that includes a morning dose for ≥ 8 weeks prior to first dose of study drug).
* BMI ≥ 25.0 kg/m2 and ≤ 40.0 kg/m2
* Additional criteria exist.

Key Exclusion Criteria:

* Recent history (i.e. less than 6 months) or concomitant/ongoing clinically significant hematologic, renal, pulmonary, gastrointestinal, hepatic, psychiatric, neurologic, dermatologic or allergic disease (including drug allergies that are clinically significant and not remote, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), or other conditions at the discretion of the investigator.
* Significant cardiac disease, myocardial infarction within 6 months of study start, unstable angina, congestive heart failure, known arrhythmias of ventricular etiology, unexplained syncope or syncope/seizures related to arrhythmia.
* History of gastric surgery, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH, or absorption.
* A positive test for drugs or alcohol.
* Active infectious diseases including hepatitis B, hepatitis C, or human immunodeficiency virus (HIV). Past history and inactive hepatitis B and C, as confirmed by serological testing, are allowed.
* Women who are pregnant or breastfeeding.
* Donation or loss of ≥ 550 mL of blood (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to first dose of study drug.
* Additional criteria exist.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, vital signs and electrocardiograms. | Duration of study
Characterize the pharmacokinetics (PK) of the study drug and metabolites in terms of plasma concentrations. | 10 days

SECONDARY OUTCOMES:
Assess the effect of study drug on glycemic control as determined by an oral glucose tolerance test (OGTT). | 10 days
Characterize the pharmacodynamic (PD) activity of the study drug on biomarkers. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Profil Institute for Clinical Research, Chula Vista, California
  - Cetero, San Antonio, Texas